CLINICAL TRIAL: NCT03703310
Title: A Multicenter, Randomized, Double-blind, Vehicle-controlled, Phase 3 Efficacy and Safety Study of Patidegib Topical Gel, 2%, for the Reduction of Disease Burden of Persistently Developing Basal Cell Carcinomas (BCCs) in Subjects With Basal Cell Nevus Syndrome
Brief Title: Study of Patidegib Topical Gel, 2%, for the Reduction of Disease Burden of Persistently Developing Basal Cell Carcinomas (BCCs) in Subjects With Basal Cell Nevus Syndrome (Gorlin Syndrome)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pelle-926-301
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2021-03

CONDITIONS: Basal Cell Nevus Syndrome
Keywords: Gorlin syndrome; Basal cell nevus syndrome BCNS; Nevoid basal cell carcinoma syndrome; Basal cell carcinoma; Hedgehog; Surgically eligible basal cell carcinomas; Patidegib
MeSH Terms: conditions — Basal Cell Nevus Syndrome; Carcinoma, Basal Cell

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to receive Patidegib Topical Gel, 2%, or Vehicle (IP)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As a double-blinded study, the Investigators, the site staff, Sponsor, and the Clinical Monitor(s) will be blinded to the treatment assigned to individual participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patidegib Topical Gel, 2%, (Experimental): Participants will be randomized to receive Patidegib Topical Gel, 2%. The Patidegib Topical Gel, 2% will be dispensed to participants at each study visit and applied topically twice daily to the face.
  Interventions: Drug: Patidegib Topical Gel, 2%
- Patidegib Topical Gel, Vehicle (Placebo Comparator): Participants will be randomized to receive Vehicle. The Patidegib Topical Gel, Vehicle will be dispensed to participants at each study visit and applied topically twice daily to the face.
  Interventions: Drug: Patidegib Topical Gel, Vehicle

INTERVENTIONS:
Drug: Patidegib Topical Gel, 2% — Patidegib Topical Gel, 2%
  Other Names: IP
  Arms: Patidegib Topical Gel, 2%,
Drug: Patidegib Topical Gel, Vehicle — Patidegib Topical Gel, Vehicle
  Other Names: IP, Vehicle
  Arms: Patidegib Topical Gel, Vehicle

SUMMARY:
This is a global, multicenter, randomized, double-blind, stratified, vehicle-controlled study of the efficacy and safety of Patidegib Topical Gel, 2%, applied topically twice daily to the face of adult participants with Gorlin syndrome. Participants will be required to apply the investigational product for 12 months. The primary endpoint is a comparison between the two treatment arms of the number of new BCCs that develop over the 12 month period.

DETAILED DESCRIPTION:
An open-label, extension safety and tolerability study is planned for at least 12 months duration following the end of this study. All participants who complete the Month 12 Exit Visit having demonstrated adequate compliance with application of the Investigational Product (IP) without major Protocol Deviations (PDs) during the study will be eligible for participation in the extension study.

All participants will be contacted by phone approximately 30 days following the Exit or Discontinuation Visit to determine if the participant has experienced any new adverse events (AEs)/serious AEs (SAEs) since discontinuation/completion of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be age at least 18 years of age at the Screening Visit.
2. The participant must provide written informed consent prior to any study procedures.
3. The participant must meet diagnostic criteria for the basal cell nevus (Gorlin) syndrome including major criterion #3a plus 1 additional major criterion or plus 2 additional minor criteria listed below.

   Major criteria:
   1. >2 histologically confirmed BCCs or 1 for participant under age 20.
   2. Odontogenic keratocysts of the jaw confirmed histologically.
   3. ≥3 palmar and/or plantar pits seen at the Screening Visit.
   4. Bilamellar calcification of the falx cerebri present at less than 20 years of age.
   5. Fused, bifid, or markedly splayed ribs.
   6. First degree relative with Gorlin syndrome.
   7. Patched protein 1 (PTCH1) mutation predicted to be of functional significance in normal tissue.

   Minor criteria:
   1. Macrocephaly.
   2. Congenital malformations including frontal bossing, cleft lip or palate, "coarse face", moderate to severe hypertelorism.
   3. Skeletal abnormalities detectable clinically: Sprengel deformity, marked pectus deformity, or marked finger syndactyly.
   4. Skeletal abnormalities detectable radiographically: bridging of the sella turcica; vertebral abnormalities such as hemivertebrae, fusion or elongation of the vertebral bodies; modeling defects of the hands and feet; flame shaped lucencies of the hands or feet.
   5. Ovarian fibroma.
   6. Medulloblastoma (Modification of criteria of V Kimonis et al Am J Med Genet 69: 299-308, 1997).
4. The participant must have 10 (with at least 3 on the face) clinically typical BCCs present within 24 months prior to Randomization (Baseline/Day 1). Additionally, the subject must have at least 2 BCCs with longest diameter <5 mm present on the face prior to Randomization (Baseline/Day 1).
5. The participant is willing to have blood collected to measure circulating drug levels.
6. The participant is willing to abstain from application of a non-study topical medication (prescription or over the counter) to facial skin for the duration of the trial except as prescribed by the Investigator. Moisturizers and emollients are allowed. Participant will be encouraged to use their preferred sunscreen with a sun protector factor (SPF) of at least 30 daily on all exposed skin sites.
7. If the participant is a woman of childbearing potential (WOCBP), she must be willing to use complete abstinence from sexual intercourse and/or she and her partner must be willing to use at least 2 highly-effective forms of birth control starting prior to Baseline, through the duration of the study, and for 12 months after last application of IP.
8. If the participant is a male with a female sex partner who is a WOCBP, the participant must be willing to use condoms, even after a vasectomy, starting prior to Baseline, through the duration of the study, and for at least 8 months after the last application of IP.
9. The participant is willing for all facial BCCs to be evaluated and treatment recommendations made only by the Investigator.
10. The participant is willing to forego treatment of facial BCCs with anything other than the study IP except when the Investigator believes that delay of treatment of a facial BCC potentially might compromise the health of the subject. During the trial the only allowed form of treatment is surgical. Non-facial BCCs may be removed at the discretion of the Investigator or Primary Skin Care Physician (PSCP).

Exclusion Criteria:

1. The subject has previously participated in a clinical trial evaluating patidegib topical gel.
2. The participant has used topical treatment to the face or systemic therapies that might interfere with the evaluation of the study IP. Among these are use of the following:

   1. 5-fluorouracil, imiquimod, diclofenac, or Ingenol mebutate (except as topical treatment to discrete non-facial BCCs) systemically or topically to the skin within the 2 months prior to the Screening Visit.
   2. Systemic chemotherapy within 1 year prior to the Screening Visit.
   3. Known inhibitors of the Hedgehog signaling pathway (such as vismodegib, sonidegib, itraconazole) topically or systemically within 3 months prior to the Screening Visit.
   4. Photodynamic therapy (PDT) except to localized non-facial, individual BCCs within 2 months prior to the Screening Visit.
3. The participant is known to have a hypersensitivity to any of the ingredients in the study medication formulation.
4. The participant is unable or unwilling to make a good faith effort to return to the study site for all study visits and tests.
5. The participant has uncontrolled systemic disease.
6. The participant has been treated for invasive cancer within the past 5 years excluding non-melanoma skin cancer, Stage I cervical cancer, ductal carcinoma in situ of the breast, or chronic lymphocytic leukemia (CLL) Stage 0.
7. The participant has current, recent (within five half-lives of the experimental drug or if half-life not known, within the past 6 months prior to the Screening Visit), or planned participation in an experimental drug study while enrolled in this study.
8. The participant is a WOCBP who is unwilling or unable to comply with pregnancy prevention measures.
9. The participant is pregnant or breastfeeding.
10. The participant has any condition or situation which, in the Investigator's opinion, may put the subject at significant risk, could confound the study results, or could interfere significantly with the subject's participation in the study. This may include a history of other skin conditions (such as severe facial eczema) or diseases, metabolic dysfunction, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the participant at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP, Clinical Operations, Study Director — PellePharm, Inc.
Locations (49):
- United States (22):
  - Mayo Clinical Cancer Center, Phoenix, Arizona
  - Dermatology Center of Newport, Newport Beach, California
  - Stanford University, Department of Dermatology, Redwood City, California
  - University of California, San Francisco, San Francisco, California
  - Yale School of Medicine, New Haven, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - Leavitt Medical Associates of Florida, Ormond Beach, Florida
  - The University of Chicago, Chicago, Illinois
  - Laser & Skin Surgery Center of Indiana, Carmel, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Dept of Dermatology, Ann Arbor, Michigan
  - University of Minnesota, Department of Dermatology, Minneapolis, Minnesota
  - Saint Louis University Dermatology, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah Midvalley Dermatology, Murray, Utah
- Belgium (2):
  - PellePharm Investigative Site, Brussels
  - PellePharm Investigative Site, Leuven
- Canada (2):
  - Clinical Trials Unit - The Skin Care Centre, Vancouver, British Columbia
  - Pellepharm Investigative Site, Toronto
- PellePharm Investigative Site, Copenhagen, Denmark
- France (6):
  - Hopital Saint-Andre - CHU Bordeaux, Bordeaux
  - CHRU de Lille - Hopital Claude HURIEZ, Lille
  - CHU La Timone, Marseille
  - PellePharm Investigative Site, Nantes
  - Hopital Saint-Louis, Paris
  - PellePharm Investigative Site, Pierre-Bénite
- Germany (4):
  - Charite - Universitatsmedizin Berlin, Berlin
  - Klinik und Poliklinik fur Dermatologie und Allergologie, Munich
  - Universitatsklinikum Münster, Münster
  - Universitats Hautklinik, Tübingen
- Italy (4):
  - Ospedale Vanvitelli-University della Campania-Dermatologia Edificio 9, Napoli
  - Catholic University of the Sacred Heart, Roma
  - Humanitas University Milan, Rozzano
  - Ospedale San Bortolo, Vicenza
- Maastricht University Medical Center - Dept of Dermatology, Maastricht, Netherlands
- Spain (3):
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitiario Virgen de la Macarena, Seville
- United Kingdom (4):
  - NHS Greater Glasgow and Clyde, Glasgow
  - Royal London Hospital, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patidegib Topical Gel, 2%, | Patidegib Topical Gel, Vehicle
Started | 87 | 87
Completed | 67 | 70
Not Completed | 20 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patidegib Topical Gel, 2%, | Patidegib Topical Gel, Vehicle | Total
Number analyzed (Participants) | 87 | 87 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (15.45) | 51.8 (13.40) | 51.8 (14.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 97
  Male | 39 | 38 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Some countries do not allow race and/or ethnicity collection
  Participants
    number analyzed (Participants) | 81 | 83 | 164
    Hispanic or Latino | 2 | 6 | 8
    Not Hispanic or Latino | 76 | 75 | 151
    Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Some countries do not allow race and/or ethnicity collection
  Participants
    number analyzed (Participants) | 82 | 84 | 166
    American Indian or Alaska Native | 0 | 2 | 2
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 79 | 78 | 157
    More than one race | 1 | 1 | 2
    Unknown or Not Reported | 2 | 3 | 5
Height [Mean (Standard Deviation); unit: cm] | 176.30 (9.390) | 176.07 (10.421) | 176.18 (9.894)
Weight [Mean (Standard Deviation); unit: kg] | 93.06 (22.812) | 91.75 (20.101) | 92.41 (21.447)
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.87 (6.062) | 29.58 (5.845) | 29.72 (5.938)
Time since Diagnosis of BCNS (basal cell nevus syndrome) [Mean (Standard Deviation); unit: years] | 28.24 (16.960) | 25.82 (16.379) | 27.03 (16.668)
Number of SEBs (surgically eligible basal cell carcinoma) at Baseline [Mean (Standard Deviation); unit: Numberof SEBs] | 4.4 (6.25) | 5.0 (6.68) | 4.7 (6.45)
Number of BCCs including SEBs at Baseline [Mean (Standard Deviation); unit: Number of BCCs] | 13.9 (11.20) | 15.4 (11.89) | 14.7 (11.54)
Number of BCCs excluding SEBs at Baseline [Mean (Standard Deviation); unit: Number of BCCs] | 9.5 (8.52) | 10.4 (8.85) | 9.9 (8.67)
Previous Hedgehog Inhibitor therapy [Number; unit: participants]
  Yes | 35 | 33 | 68
  No | 52 | 54 | 106

OUTCOME MEASURES:

1. Primary Outcome: Number of New BCCs Per Participant
Time Frame: Month 12
Population: The number of BCCs per subject by Month 12 summarized subjects with BCC assessments within the Month 12 analysis window.
Measure: Mean (Standard Deviation); unit: New basal cell carcinomas
Arm/Group | Patidegib Topical Gel, 2%, | Patidegib Topical Gel, Vehicle
Number analyzed (Participants) | 58 | 65
New basal cell carcinomas | 2.84 (3.39) | 4.03 (4.76)

2. Secondary Outcome: Number of New Surgically Eligible BCCs (nSEBs) Per Participant
Time Frame: Month 12
Population: The number of nSEBs per subject by Month 12 summarizes subjects with BCC assessments within the Month 12 analysis window.
Measure: Mean (Standard Deviation); unit: New basal cell carcinomas
Arm/Group | Patidegib Topical Gel, 2%, | Patidegib Topical Gel, Vehicle
Number analyzed (Participants) | 58 | 65
New basal cell carcinomas | 0.71 (1.28) | 0.91 (1.61)

3. Secondary Outcome: Percentage of Participants Developing >=2 Facial New BCCs
Time Frame: Month 12
Population: subjects with no postbaseline data were excluded from the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Patidegib Topical Gel, 2%, | Patidegib Topical Gel, Vehicle
Number analyzed (Participants) | 83 | 86
Participants | 45 | 55

4. Secondary Outcome: Percentage of Participants Developing >=1 Facial New BCCs
Time Frame: Month 12
Population: subjects with no postbaseline data were excluded from the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Patidegib Topical Gel, 2%, | Patidegib Topical Gel, Vehicle
Number analyzed (Participants) | 83 | 86
Participants | 56 | 65

5. Secondary Outcome: Number of New BCCs Per Participant
Time Frame: Month 9
Population: subjects with no postbaseline data were excluded from the analysis
Measure: Mean (Standard Deviation); unit: New basal cell carcinomas
Arm/Group | Patidegib Topical Gel, 2%, | Patidegib Topical Gel, Vehicle
Number analyzed (Participants) | 68 | 65
New basal cell carcinomas | 2.46 (3.42) | 3.15 (3.94)

6. Secondary Outcome: Number of New BCCs Per Participant
Time Frame: Month 6
Population: subjects with no postbaseline data were excluded from the analysis
Measure: Mean (Standard Deviation); unit: New basal cell carcinomas
Arm/Group | Patidegib Topical Gel, 2%, | Patidegib Topical Gel, Vehicle
Number analyzed (Participants) | 68 | 69
New basal cell carcinomas | 1.68 (2.82) | 2.12 (2.96)

7. Secondary Outcome: Change in Advanced Basal Cell Carcinoma Index (aBCCdex) Lesion Symptom Score Scale Score
Description: The Advanced Basal Cell Carcinoma Index (aBCCdex) measures the impact of basal cell carcinoma on patients' quality of life. The index consists of several subscales, each subscale with its own range of scores for each question
  Lesion Symptoms Scale: Scores range from 1 to 7 and it includes 6 questions. Therefore the total score range is from 6 (minimum) to 42 (maximum), where a higher score correlates with a poorer quality of life.
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patidegib Topical Gel, 2%, | Patidegib Topical Gel, Vehicle
Number analyzed (Participants) | 87 | 87
score on a scale | 11.49 (18.365) | 15.54 (21.002)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Patidegib Topical Gel, 2%, | Patidegib Topical Gel, Vehicle
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/87
Serious Adverse Events (participants affected / at risk) | 5/87 | 7/87
Other Adverse Events (participants affected / at risk) | 47/87 | 65/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patidegib Topical Gel, 2%, (N=87) | Patidegib Topical Gel, Vehicle (N=87)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Vaginal abscess (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Morton's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patidegib Topical Gel, 2%, (N=87) | Patidegib Topical Gel, Vehicle (N=87)
Upper respiratory tract infection (Infections and infestations) | 5 | 9
Urinary tract infection (Infections and infestations) | 5 | 6
Nasopharyngitis (Infections and infestations) | 2 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 9
Fatigue (General disorders) | 5 | 4
Pyrexia (General disorders) | 5 | 1
Headache (Nervous system disorders) | 5 | 8
Paraesthesia (Nervous system disorders) | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT03703310/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT03703310/SAP_001.pdf